CLINICAL TRIAL: NCT01867125
Title: A Phase III, Randomized, Double-Blind, Placebo-Controlled Study to Assess the Efficacy and Safety of Lebrikizumab in Patients With Uncontrolled Asthma Who Are on Inhaled Corticosteroids and a Second Controller Medication
Brief Title: A Study of Lebrikizumab in Participants With Uncontrolled Asthma Who Are on Inhaled Corticosteroids and a Second Controller Medication
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GB28688; 2013-000175-33 (EudraCT Number)
Record Dates: First submitted 2013-05-29; First posted 2013-06-03 (Estimated); Last update posted 2017-05-19 (Actual); Status verified 2017-05

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — lebrikizumab

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Lebrikizumab (125 mg) (Experimental): Participants will receive SC injection of lebrikizumab (125 milligrams [mg]) every 4 weeks for 104 weeks.
  Interventions: Drug: Lebrikizumab
- Lebrikizumab (37.5 mg) (Experimental): Participants will receive SC injection of lebrikizumab (37.5 mg) every 4 weeks for 104 weeks.
  Interventions: Drug: Lebrikizumab; Drug: Placebo
- Placebo (Placebo Comparator): Participants will receive SC injection of lebrikizumab matching placebo every 4 weeks for 52 weeks during placebo-controlled period and then SC injection of lebrikizumab at 125 or 37.5 mg for 52 weeks during active treatment extension period.
  Interventions: Drug: Lebrikizumab; Drug: Placebo

INTERVENTIONS:
Drug: Lebrikizumab — Lebrikizumab will be administered as SC injection at 125 or 37.5 mg every 4 weeks, for 104 weeks.
  Other Names: RO5490255
Drug: Placebo — Lebrikizumab matching placebo will be administered as SC injection every 4 weeks for 52 weeks.
  Arms: Lebrikizumab (37.5 mg); Placebo

SUMMARY:
This randomized, multicenter, double-blind, placebo-controlled, parallel-group study will evaluate the efficacy and safety of lebrikizumab in participants with asthma whose disease remains uncontrolled despite daily treatment with inhaled corticosteroid (ICS) therapy and at least one second controller medication. Participants will be randomized in 1:1:1 ratio to receive double-blind treatment with either lebrikizumab ("high" or "low") or placebo, administered subcutaneously (SC) every 4 weeks for 52 weeks, in addition to their standard-of-care therapy. This will be followed by a 52-week double-blind active treatment extension. During double-blind active treatment extension period, all participants will receive SC injection of lebrikizumab from Week 53 to Week 104. The anticipated time on study treatment is 104 weeks. After study treatment, all participants will complete a 20-week safety follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Asthma diagnosis for greater than equal to (>/=) 12 months prior to Visit 1
* Bronchodilator response at Visit 1, 2, or 3
* Pre-bronchodilator FEV1 of 40 percent (%) - 80% predicted at both Visits 2 and 3
* On ICS therapy at a total daily dose of 500-2000 micrograms (mcg) of fluticasone propionate dry powder inhaler (DPI) or equivalent for >/=6 months prior to Visit 1
* On an eligible second controller medication (long-acting beta-agonist [LABA], leukotriene receptor antagonist [LTRA], long-acting muscarinic antagonist [LAMA], or theophylline) for 6 months prior to Visit 1
* Uncontrolled asthma at Visit 1 and/or Visit 2, and at Visit 3
* Chest X-ray or computed tomography (CT) scan within 3 months prior to Visit 1 or chest X-ray during the screening period (prior to Visit 3) confirming the absence of other clinically significant lung disease
* Demonstrated adherence with controller medication during the screening period

Exclusion Criteria:

* History of severe allergic reaction or anaphylactic reaction to a biologic agent or known hypersensitivity to any component of the lebrikizumab injection
* Maintenance oral corticosteroid therapy within 3 months of Visit 1
* Treatment with systemic (oral, intravenous [IV], or intramuscular [IM]) corticosteroids within 4 weeks prior to Visit 1 or during the screening period
* Treatment with intra-articular corticosteroids within 4 weeks prior to Visit 1 or during the screening period or anticipated need for intra-articular corticosteroids during the course of the study
* Infection requiring hospital admission for >/=24 hours or requiring treatment with IV or IM antibiotics within 4 weeks prior to Visit 1 or during screening; Upper or lower respiratory tract infection within 4 weeks prior to Visit 1 or during screening; Active infection that required treatment with oral antibiotics within 2 weeks prior to Visit 1 or during screening; Active parasitic infection or Listeria monocytogenes infection within 6 months prior to Visit 1 or during screening
* Active tuberculosis requiring treatment within 12 months prior to Visit 1
* Known immunodeficiency, including, but not limited to, human immunodeficiency virus (HIV) infection
* Evidence of acute or chronic hepatitis or known liver cirrhosis
* History of interstitial lung disease, chronic obstructive pulmonary disease (COPD), or other clinically significant lung disease other than asthma
* Known current malignancy or current evaluation for potential malignancy
* Current smoker or former smoker with a history of greater than (>) 10 pack-years
* History of alcohol or drug abuse
* Past and/or current use of any anti-interleukin (IL)-13 or anti-IL-4/IL-13 therapy, including lebrikizumab
* Use of other monoclonal antibody therapy, including omalizumab, within 6 months or 5 drug half-lives prior to Visit 1 (whichever is longer) or during screening
* Initiation of or change in allergen immunotherapy within 3 months prior to Visit 1 or during screening

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1081 (Actual)
Dates: Start 2013-07-31 (Actual); Primary Completion 2017-01-02 (Actual); Study Completion 2017-01-02 (Actual)

PRIMARY OUTCOMES:
Rate of Asthma Exacerbations During the 52-Week Placebo-Controlled Period | Baseline up to 52 weeks

SECONDARY OUTCOMES:
Absolute Change From Baseline in Pre-Bronchodilator Forced Expiratory Volume in 1 Second (FEV1) | Baseline, Week 52
Time to First Asthma Exacerbation | Baseline up to 52 weeks
Change From Baseline in Standardized Asthma Quality of Life Questionnaire (AQLQ) Score | Baseline, Week 52
Change from Baseline In Asthma Rescue Medication (Number of Puffs or Nebulized Treatments) | Baseline, Week 52
Rate of Urgent Asthma-Related Urgent Health Care Utilization | Baseline up to Week 52
Percentage of Participants With Anti-Therapeutic Antibodies to Lebrikizumab | Baseline up to Week 124 (assessed at Baseline, Weeks 4, 12, 24, 36, 52, 64, 76, 92, 104, 112, and 124)
Change From Baseline in Asthma Control Questionnaire-5 (ACQ-5) Score | Baseline, Week 52
Percentage of Participants With Adverse Events | Baseline, Week 124
Minimum Serum Concentration (Cmin) of Lebrikizumab | Predose (0 hour) on Weeks 4, 12, 24, 36, and 52

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (230):
- United States (69):
  - Alabama Clinical Research Associates, Pell City, Alabama
  - Clinical Trial Connection, Flagstaff, Arizona
  - Desert Sun Clinical Research LLC, Tucson, Arizona
  - Allianz Medical and Research Center, Fountain Valley, California
  - Allergy & Asthma Medical Group & Research Center, Pc, Long Beach, California
  - Alliance Research LLC, Long Beach, California
  - Allergy Medical Clinic, Los Angeles, California
  - CA Allergy & Asthma Med Grp, Los Angeles, California
  - North Bay Clinical Trials, Napa, California
  - Choc Psf, Amc, Orange, California
  - Advances in Medicine, Rancho Mirage, California
  - Allergy Assoc Medical Group, San Diego, California
  - UCSF School of Medicine, San Francisco, California
  - Bensch Research Associates, Stockton, California
  - IMMUNOe International Research Centers, Centennial, Colorado
  - Waterbury Pulmonary Associates, Waterbury, Connecticut
  - St. Francis Sleep; Allergy & Lung Institute, Clearwater, Florida
  - Creekside Medical Research, DeLand, Florida
  - Suncoast Research Group LLC, Miami, Florida
  - South Florida Research Phase I-IV, Inc, Miami, Florida
  - Allergy & Asthma Care of FL; Clinical Research, Ocala, Florida
  - Emerald Coast Research Associates, Panama City, Florida
  - Allergy & Asthma Diagnostic; Treatment Center, Tallahassee, Florida
  - Florida Pulmonary Research Institute, LLC, Winter Park, Florida
  - Southeastern Lung Care, Decatur, Georgia
  - Atlanta Allergy & Asthma Clini, Woodstock, Georgia
  - Laporte County Institute For Clinical Research, Michigan City, Indiana
  - Iowa Clinical Research Corporation, Iowa City, Iowa
  - Northeast Medical Research Associates, Inc, North Dartmouth, Massachusetts
  - Infusion Associates, Grand Rapids, Michigan
  - Midwest Clinical Research LLC, St Louis, Missouri
  - Washington Univ. School of Med, St Louis, Missouri
  - Montana Medical Research LLC, Missoula, Montana
  - Heartland Clinical Research Inc., Omaha, Nebraska
  - Asthma & Allergy Center, P.C., Papillion, Nebraska
  - Allergy & Asthma Associates, Las Vegas, Nevada
  - Allergy & Asthma Research of Nj, Inc, Mount Laurel, New Jersey
  - Atlantic Research Center, LLC, Ocean City, New Jersey
  - Princeton Center For Clinical Research, Skillman, New Jersey
  - North Shore University Hosp, New Hyde Park, New York
  - Montefiore Medical Center, The Bronx, New York
  - Allergy & Asthma Center of NC, High Point, North Carolina
  - PMG Research of Wilmington, Wilmington, North Carolina
  - Asthma & Allergy Center, Toledo, Ohio
  - Cor Clinical Research, Oklahoma City, Oklahoma
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Allergy & Asthma Research Grp, Eugene, Oregon
  - Clinical Research Inst. of Southern Oregon, Pc, Medford, Oregon
  - Allergy Associates Research Center, Portland, Oregon
  - Central PA Asth & Allergy Care; Research Division, Altoona, Pennsylvania
  - Asthma Allergy Pulm Associates, Philadelphia, Pennsylvania
  - Grand View Hospital; Clinical Research Department, Sellersville, Pennsylvania
  - Asthma Allergy Phys of RI, Lincoln, Rhode Island
  - ADAC Research PA, Greenville, South Carolina
  - Spartanburg Medical Research, Spartanburg, South Carolina
  - Tekton Research Inc, Austin, Texas
  - TTS Research, Boerne, Texas
  - Pharmaceutical Research & Consulting, Inc., Dallas, Texas
  - Allergy & Asthma Research Center of El Paso, El Paso, Texas
  - Pioneer Research Solutions, Houston, Texas
  - Metroplex Pulmonology & Sleep Center, McKinney, Texas
  - Quality Assurance Research Ctr, San Antonio, Texas
  - O & O Alpan, LLC, Fairfax, Virginia
  - Clinical Research Partners, LLC, Henrico, Virginia
  - Manassas Clinical Research Center, Manassas, Virginia
  - Bellingham Asthma, Allergy & Immunology, Bellingham, Washington
  - ASTHMA, Inc, Seattle, Washington
  - Marycliff Allergy Specialists, Spokane, Washington
  - Dean Clinic, Madison, Wisconsin
- Argentina (5):
  - Fundación Faicep, Buenos Aires
  - Centro Médico Dra de Salvo, Buenos Aires
  - Instituto Ave Pulmo, Mar del Plata
  - Centro Respiratorio Quilmes, Quilmes
  - Investigaciones en Patologias Respiratorias, San Miguel de Tucumán
- Australia (5):
  - Liverpool Hospital, Liverpool BC, New South Wales
  - St. Vincent's Hospital Melbourne, Fitzroy, South Australia
  - Box Hill Hospital; Eastern Clinical Research Unit, Box Hill, Victoria
  - Western Hospital, Footscray, Victoria
  - The Lung Institute of Western Australia; Sir Charles Gairdner Hospital, Nedlands, Western Australia
- Belgium (2):
  - Cliniques Universitaires St-Luc, Brussels
  - UZ Gent, Ghent
- Canada (5):
  - Alberta Health Services, Calgary, Alberta
  - Dr. E. Amer, Mississauga, Ontario
  - Inspiration Research Limited, Toronto, Ontario
  - Albion Finch Medical Centre, Toronto, Ontario
  - Centre d'investigation Clinique Mauricie, Trois-Rivières, Quebec
- Chile (3):
  - Centro de Investigaciones Medicas Respiratorias, Santiago
  - Schonffeldt y Guerrero Limitada, Santiago
  - Hospital Carlos Van Buren, Valparaíso
- Fundacion Neumologica Colombiana, Bogota DC, Colombia
- Czechia (4):
  - Alergopraktik s.r.o., Jablonec nad Nisou
  - Interni A Pneumologicka Ambulance, Jindřichův Hradec
  - MephaCentrum, a.s., Ostrava - Poruba
  - Alergologie Teplice, s.r.o., Teplice
- France (5):
  - Hopital Calmette; Pneumologie, Lille
  - Hopital Nord; CIC, Marseille
  - Hôpital Arnaud de Villeneuve, Montpellier
  - CHU Nantes - Hôpital Laennec; Service de Pneumologie, Nantes
  - Nouvel Hôpital Civil; Pôle de Pathologie Thoracique, Strabourg
- Germany (2):
  - Lungenarztpraxis Tegel, Berlin
  - Pneumologisches Zentrum Wiesloch, Wiesloch
- Hungary (3):
  - Kenezy Korhaz Rendelointezet, Debrecen
  - Petz Aladar Megyei Oktato Korhaz, Győr
  - C.C.C. Hospital Chest Diseases, Szeged
- Israel (5):
  - Barzilai Medical Center; Pulmonary Inst., Ashkelon
  - Lady Davis Carmel Medical Center; Cardiovascular Medicine, Haifa
  - Shaare Zedek Medical Center, Jerusalem
  - Meir Medical Center; Pulmonary Dept, Kfar Saba
  - Kaplan Medical Center, Rehovot
- Italy (6):
  - Fondazione Salvatore Maugeri. IRCCS - Divisione di Pneumologia, Cassano Murge (BA), Apulia
  - University of Catanzaro, Catanzaro, Calabria
  - Azienda Ospedaliero Universitaria di Parma, Parma, Emilia-Romagna
  - Azienda Ospedaliero Universitaria Ospedali Riuniti Umberto I-G.M. Lancisi-G. Salesi Di Ancona, Torrette - Ancona, The Marches
  - A.o. Universitaria Pisana; Dipartimento Cardio Toracico, Pisa, Tuscany
  - Azienda Ospedaliera di Padova, Padua, Veneto
- Japan (29):
  - Tosei General Hospital; Respiratory and Allergy Medicine, Aichi
  - Ofuji Clinic, Amagasaki-shi
  - Kyushu Central Hospital, Fukuoka
  - National Hospital Organization Mito Medical Center, Higashiibaraki-gun
  - Hiroshima University Hospital, Hiroshima
  - Oji General Hospital, Hokkaido
  - National Hospital Organization Asahikawa Medical Center, Hokkaido
  - Yokohama City Minato Red Cross Hospital, Kanagawa
  - National Hospital Organization Tokyo National Hospital, Kiyose-shi
  - Kochi Medical School Hospital, Kochi
  - Oki Clinic, Kodaira-shi
  - Takahashi Clinic, Kokubunji-shi
  - Dokkyo Medical University Koshigaya Hospital, Koshigaya-shi
  - Tono Chuo Clinic, Mizunami-shi
  - Nagaoka Red Cross Hospital, Nagaoka-shi
  - Niigata City General Hospital, Niigata
  - Iwate Medical University Hospital, Numakunai
  - Osaka City University Hospital, Osaka
  - Touda Clinic, Osaka
  - Kinki-Chuo Chest Medical Center, Osaka
  - Senzoku Kokyuuki and Allergy Clinic, Ōta-ku
  - Japan Community Health Care Organization Hokkaido Hospital, Sapporo
  - Fukuwa Clinic, Tokyo
  - Tokyo Center Clinic; Internal Medicine, Tokyo
  - Sano Toranomon Clinic, Tokyo
  - Showa University Hospital, Tokyo
  - Teikyo University Hospital, Tokyo
  - Sekino Hospital, Toshima City
  - University of Fukui Hospital, Yoshida-gun
- Mexico (2):
  - Instituto Jalisciense de Investigacion Clinica S.A. de C.V., Guadalajara
  - Hospital Dr Angel Leaño universidad Autonoma de Guadalajara AC, Zapopan
- New Zealand (4):
  - NZ Respiratory & Sleep Institute, Auckland
  - Dunedin Hospital, Dunedin
  - RMC Medical Research Ltd, Dunedin
  - P3 Research, Tauranga
- Poland (12):
  - Centrum Medycyny Oddechowej Robert M. Mróz, Bialystok
  - Prywatna Praktyka Lekarska Gabinet Pediatryczno-Alergologiczny, Bialystok
  - Specjalistyczne Centrum Medyczne NOWOMED, Krakow
  - Grazyna Pulka Specjalistyczny Ośrodek ALL-MED, Krakow
  - Niepubliczny Zaklad Opieki Zdrowotnej Centrum Medyczne ProMiMed sp z o.o. sp.k., Krakow
  - Poradnia Pulmonologiczna dla Doroslych, Lódz
  - Centrum Alergologii Teresa Hofman, Poznan
  - SPZOZ Proszowice, Proszowice
  - Niepubliczny Specjalistyczny ZOZ Puls-Med s.c., Skarżysko-Kamienna
  - Medica Pro Familia Sp. z o.o. S.K.A., Warsaw
  - Klinika Chorób Wewnetrznych i Alergologii MSW, Warsaw
  - ALL-MED Specjalistyczna Opieka Medyczna, Wroclaw
- Romania (4):
  - Colentina Clinical Hospital, Bucharest
  - Prof.Dr.Octavian Fodor Emergency Clinical Hospital, Cluj-Napoca
  - Spitalul Clinic de Boli Infectioase si Pneumoftiziologie Victor Babes Craiova, Craiova
  - Dr. Victor Babes Pneumology and Infectious Diseases Clinical Hospital, Timișoara
- Russia (13):
  - SIH Kemerovo Regional Clinical Hospital, Kemerovo
  - Russian Uni of People'S Friendship, Med. Faculty; City Clinical Hospital No 64, Internal Diseases, Moscow
  - Central Clinical Hospital #1 of RZhD JCS, Moscow
  - Novosibirsk Municipal Clinical Hospital For Emergency Medicine #2, Novosibirsk
  - Ryazan Regional Clinical Hosp, Ryazan
  - City Outpatient Dept #94, Saint Petersburg
  - St-Petersburg Diagnostic Ctr#1; Pulmonology, Saint Petersburg
  - SHI Ctr Occupational Pathology, Saint Petersburg
  - St. Petersburg State Budget Medical Institution Pokrovskaya City Hospital, Saint Petersburg
  - St.-Petersburg SMU n. a. Academician I.P.Pavlov; Therapy Department, Saint Petersburg
  - St. George the Martyr City Hospital, Saint Petersburg
  - Smolensk State Medical Academy, Smolensk
  - Tomsk Regional Clinical Hospital, Tomsk
- Serbia (3):
  - Clinical Center of Serbia, Belgrade
  - Clinical Hospital Center Zvezdara, Belgrade
  - Clinical Hospital Center ''Bezanijska Kosa''; Department of Pulmology, Belgrade
- Slovakia (3):
  - Alian s.r.o., Bardejov
  - Tehelná Clinic, Inc; IMUNO-ALERGO, s. r.o., Bratislava
  - Plucna ambulancia, Spišská Nová Ves
- South Africa (7):
  - Melomed Hospital Gatesville, Cape Town
  - Uni of Cape Town Lung Inst., Cape Town
  - Vawda Z.Fa Practice, Durban
  - Gatesville Medical Centre, Gatesville
  - Deepak Lakha MBCHB Private Practice, Johannesburg
  - Botho ke Bontle Health Services, Pretoria
  - Dr Johannes Breedt; Emmed Research, Pretoria
- South Korea (6):
  - Seoul National University Bundang Hospital, Gyeonggi-do
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Korea University Guro Hospital, Seoul
  - St. Paul's Hospital, The Catholic University of Korea, College of Medicine, Seoul
  - Wonju Christian Hospital, Wŏnju
- Spain (6):
  - Hospital Universitario Araba, Vitoria-Gasteiz, Alava
  - Hospital de la Santa Creu; i Sant Pau, Barcelona
  - Hospital Germans Trias i Pujol, Barcelona
  - Hosp Univ Fundacion Alcorcon, Madrid
  - Hospital Virgen del Rocio, Seville
  - Hospital Universitario Doctor Peset, Valencia
- Turkey (Türkiye) (8):
  - Atatürk Göğüs Hastalıkları ve Göğüs Cerrahisi Eğitim ve Araştırma Hastanesi, Ankara
  - Turgut Ozal Universitesi Tip Fakultesi Bestepe Hastanesi, Ankara
  - Uludag University; Pulmonology and Allergy Department, Bursa
  - Canakkale Onsekiz Mart Universitesi Tip Fakultesi Hastanesi, Çanakkale
  - Ege University Medical Faculty, Izmir
  - Izmir Dr. Suat Seren Gogus Hastaliklari ve Cerrahisi Egitim ve Arastirma Hastanesi, Izmir
  - Kirikkale Universitesi Tip Fakultesi Hastanesi, Kırıkkale
  - Mersin University Medical Faculty, Mersin
- Ukraine (13):
  - Public Institution City Clinical Hospital # 6 of Dnipropetrovsk Regional Board, Dnipro
  - Educational Scientific Medical Centre of Donetsk National Medical University;, Donetsk
  - Regional Phthisiology and Pulmonology Center, Ivano-Frankivsk
  - City Clinical Hospital #27, Kharkiv
  - Medical and Sanitary Unit of OJSC "Kharkiv Tractor Plant n.a. Ordzhonikidze"; Department of Therapy, Kharkiv
  - Central Outpatient Hospital of Desnyansky District, Kyiv
  - Yanovskyy Inst of Phth. & Pulm; Clinical-functional, Kyiv
  - Municipal Institution of Kyiv Regional Council Kyiv Regional Clinical Hospital, Kyiv
  - Kyiv City Clinical Hospital #8, Kyiv
  - Danylo Halytskyy National Medical University; Lviv, Lviv
  - Small Business Private Enterprise Medical Centre Pulse, Vinnytsia
  - Municipal Institution of Health Care "Yevpatoriya City Hospital №1, Yevpatoria
  - SI Dept. Clin. Hospital of Zaporizhzhia-2 Railway Station of SE Prydniprovska Zaliznytsia, Zaporizhzhia
- United Kingdom (5):
  - St Peters Hospital, Chertsey
  - Castle Hill Hospital; Respiratory Medicine, Cottingham
  - Ninewells Hospital; Asthma and Allergy Research Group, Dundee
  - St James University Hospital; Respiratory Department, Leeds
  - University North Tees, Teesside

REFERENCES:
- [Derived] Chen M, Shepard K 2nd, Yang M, Raut P, Pazwash H, Holweg CTJ, Choo E. Overlap of allergic, eosinophilic and type 2 inflammatory subtypes in moderate-to-severe asthma. Clin Exp Allergy. 2021 Apr;51(4):546-555. doi: 10.1111/cea.13790. Epub 2021 Jan 7. PMID 33217063
- [Derived] N Bauer R, Yang X, L Staton T, Olsson J, Holweg CTJ, R Arron J, Matthews JG, Choy DF. Seasonal variability of lung function and Asthma Quality of Life Questionnaire Scores in adults with uncontrolled asthma. BMJ Open Respir Res. 2019 Nov 11;6(1):e000406. doi: 10.1136/bmjresp-2019-000406. eCollection 2019. PMID 31803473
- [Derived] Hanania NA, Korenblat P, Chapman KR, Bateman ED, Kopecky P, Paggiaro P, Yokoyama A, Olsson J, Gray S, Holweg CT, Eisner M, Asare C, Fischer SK, Peng K, Putnam WS, Matthews JG. Efficacy and safety of lebrikizumab in patients with uncontrolled asthma (LAVOLTA I and LAVOLTA II): replicate, phase 3, randomised, double-blind, placebo-controlled trials. Lancet Respir Med. 2016 Oct;4(10):781-796. doi: 10.1016/S2213-2600(16)30265-X. Epub 2016 Sep 5. PMID 27616196